CLINICAL TRIAL: NCT07144072
Title: A Phase I, Open-Label, Dose-Escalation Study to Evaluate the Safety and Tolerability of HeXell-2020 Administered Intravenously in Elderly Subjects With Mild to Moderate Frailty Syndrome
Brief Title: Safety and Tolerability Study of Mesenchymal Stem Cells, HeXell-2020, in Elderly Subjects With Mild to Moderate Frailty Syndrome
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hexun Biosciences Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HeXell-2020-FS-001
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Frailty in Older Adults
Keywords: HeXell-2020; Mesenchymal Stem Cells (MSC); Frailty Syndrome (FS)
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Single arm, 2 dose cohorts with dose-defining escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cell Drug:HeXell-2020 (Experimental): Two cohort. Cohort 1: HeXell-2020 will be administered by intravenous once every two weeks, and a total of 3 doses.
  Cohort 2: HeXell-2020 will be administered by intravenous once every two weeks, and a total of 6 doses.
  Interventions: Drug: HeXell-2020

INTERVENTIONS:
Drug: HeXell-2020 — Cohort 1: 5 × 10⁷ cells per dose, administered via IV infusion every 2 weeks for a total of 3 doses Cohort 2 : 5 × 10⁷ cells per dose, administered via IV infusion every 2 weeks for a total of 6 doses

SUMMARY:
This is a phase I study to investigate the safety, and Tolerability of HeXell-2020 in Elderly Subjects with Mild to Moderate Frailty Syndrome.

HeXell-2020 is an investigational drug product consisting of allogenic umbilical cord mesenchymal stem cells (UCMSCs) as the drug substance. All enrolled and eligible subjects will receive HeXell-2020 treatment.

DETAILED DESCRIPTION:
Frailty Syndrome (FS) is a complex clinical phenotype characterized by increased vulnerability and reduced physiological reserve resulting from progressive decline across multiple physiological systems. Clinically, FS is manifested by reduced grip strength, exhaustion, slower walking speed, low physical activity, and unintentional weight loss. This condition is associated with elevated oxidative stress, chronic inflammation, decreased muscle mass, and organ dysfunction, which collectively contribute to an increased risk of disability, hospitalization, and mortality.

The pharmacological efficacy of MSCs has been extensively investigated including the secretion of immunomodulatory molecules, antioxidative enzymes, pro-angiogenic growth factors, and anti-apoptotic agents that collectively target multiple pathological mechanisms underlying frailty syndrome. UC-MSCs also exert potent anti-apoptotic effects by upregulating the expression of anti-apoptotic protein and simultaneously downregulating cellular senescence and apoptosis.

The investigational Drug Product (DP), HeXell-2020, consists of allogeneic umbilical cord-derived mesenchymal stem cells (UC-MSCs) isolated from human Wharton's jelly, which is intended to treat patients with FS. A GLP-compliant eleven repeated-dose (once every 7 days) toxicity study (Study Number 21005IV01), in which three does levels (1.5 × 10e6, 1.5 × 10⁷, 7.5 × 10⁷ cells/kg/dose) of HeXell-2020 or vehicle control was administered to NOD/SCID mice, was conducted to evaluate toxicity, local tolerance, and biodistribution. During the observation period, most of the survived animals appeared normal in all control and treated groups after dosing. The MTD (maximum tolerated dose) of HeXell-2020 is determined to be 1.5 × 10⁷ cells/kg/dose for 11 doses.

In current in vivo studies, rodents were administered UC-MSCs, which effectively restored skeletal muscle function by modulating extracellular matrix composition, activating muscle satellite cells, promoting autophagy, and mitigating cellular senescence through down-regulation of intracellular senescence signaling pathways. These mechanisms led to improved muscle mass, strength, and physical performance, directly addressing core symptoms of frailty. MSCs were observed to promote angiogenesis and improve tissue perfusion by secreting angiogenic factors, thereby facilitating capillary network formation and accelerating tissue regeneration.

This is a Phase I, open-label, dose-escalation study designed to evaluate the safety and tolerability of HeXell-2020 in elderly subjects with mild to moderate FS. Subjects aged 60 to 85 years will be enrolled. Up to 12 subjects will be sequentially allocated, and the study will follow a standard "3+3" dose-escalation design to determine the Maximum Feasible Dose (MFD). This study is designed to evaluate the safety of human umbilical cord-derived mesenchymal stem cells (UC-MSCs) product HeXell-2020 intravenous infusion in frail adults prior to further clinical development.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet ALL the following criteria at time of Screening:

1. Subjects aged ≥ 60 through ≤ 85 years old.
2. Subjects with clinical diagnosis of mild to moderate Frailty Syndrome as assessed by the Investigator with a Clinical Frailty Scale score between 4 to 6.
3. Subject will not start any new treatment for this condition during the study.
4. Subjects with body weight between 40 to 90 kg.
5. Subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided.

Exclusion Criteria:

Subjects meeting ANY of the following criteria at time of Screening will be excluded from enrollment:

1. Subjects unwilling or unable to perform any of the assessments required by endpoint analysis.
2. Subjects who have a diagnosis of any disabling neurologic disorder including, but not limited to: Parkinson's disease, Amyotrophic Lateral Sclerosis, multiple sclerosis, stroke or dementia.
3. Subjects who have a score on the Mini-Mental State Examination (MMSE) of 24 or below.
4. Subjects who have a significant comorbid medical condition(s) including, but not limited to:

   1. Severe kidney disease requiring hemodialysis or peritoneal dialysis;
   2. Advanced liver disease such as severe liver cirrhosis;
   3. Severe congestive heart failure (NYHA class 3 and 4);
   4. Severe pulmonary dysfunction, including severe chronic obstructive pulmonary disease stage III or IV (Gold classification)
5. Subjects who have a clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease free for 5 years), except curatively-treated basal cell carcinoma or in situ carcinomas.
6. Subjects using chronic immunosuppressant therapy, including corticosteroids (> 5 mg/day of prednisone, or equivalent), or TNF-alpha antagonists.
7. Subjects on chronic immunosuppressive transplant therapy.
8. Subjects who have participated in another clinical study of new investigational therapies within 6 months prior to screening.
9. Subjects who have received any other stem cell therapy within 12 months prior to screening.
10. Subjects with known allergy or hypersensitivity to any component of the formulation and cellular therapies (i.e., penicillin or streptomycin).
11. Subjects who have a history of drug or alcohol abuse within the past 3 years.
12. Subjects who are known to be infected with HIV.
13. Subjects currently in hospital stay.
14. Subjects who have a significant illness as judged by principal investigator (PI) including, but not limited to:

    1. Psychiatric illness
    2. Uncontrolled hypertension or hypotension
    3. Unstable cardiac arrhythmia
    4. Active Hepatitis B, Hepatitis C infections
15. Subjects who have any condition that in the opinion of the Principal Investigator limits lifespan to < 1 year.
16. Subjects who have any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Feasible Dose (MFD) determination | Within 14 days after completion of the last study treatment (day 28 for 3 doses treatment and day 70 for 6 doses treatment ) .
  MFD is determined on the occurrence of Dose Limiting Toxicities (DLTs) after IV administration in elderly subjects with mild to moderate FS. DLT is defined as any clinically significant adverse event (AE)/serious adverse event (SAE) or clinically significant laboratory abnormality which is classified as ≥ Grade 3 (according to the National Cancer Institute Common Terminology Criteria for Adverse Events [CTCAE] version 5.0), where applicable, is assessed as unrelated to disease progression, concurrent illness, or concomitant medications and occurring within 14 days after completion of the last study treatment .
Incidence of Treatment-Emergent Adverse Events (TEAEs). | Within the first year after cell transplantation.
  TEAE are defined as adverse events with onset date on or after the first treatment. TEAEs will be summarized by treatment group, System Organ Class, and preferred term. The following TEAE summaries will be provided:
  1. Overall (i.e., regardless of severity or relationship to treatment)
  2. Adverse events by severity
  3. Related adverse events by severity
  4. Adverse events leading to treatment discontinuation by severity
  5. Adverse events leading to death by severity
Incidence of withdrawals due to AEs | Within the first year after cell transplantation.
  An adverse event (AE) is will be classified by system organ class (SOC) and preferred term (PT) according to the most recent version of MedDAR dictionary.

SECONDARY OUTCOMES:
Mean change from baseline in exercise performance as measured by change in the six-minute walk test (6MWT) total distance. | Day 0 (baseline), Week 6, 12, 24, 36, 52
  The six-minute walk test (6MWT) measures the total distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Mean change from baseline in hand grip strength as measured by change in maximum force using hand dynamometer. | Day 0 (baseline), Week 6, 12, 24, 36, 52
  Hand grip strength is a measure of the maximum static force that a hand can squeeze using a Baseline Hydraulic Hand Dynamometer.
Mean change from baseline in physical activity as measured by change in the Short Physical Performance Battery (SPPB) assessment total score. | Day 0 (baseline), Week 6, 12, 24, 36, 52
  The Short Physical Performance Battery (SPPB) Total Score is a measure of physical function. It is calculated by summing three measures of lower-extremity function: standing balance (side-by-side, semi-tandem, and tandem stance), 4-meter walking speed, and ability to rise from a chair. Each task is rated on a 0-4 scale, with increasing scores indicating better physical performance. The SPPB Total scores range from 0-12.
Mean change from baseline in Clinical Frailty Scale (CFS) score. | Day 0 (baseline), Week 6, 12, 24, 36, 52
  The Clinical Frailty Scale (CFS) is a common way to summarize the overall level of fitness or frailty of an elderly after they had been evaluated by an experienced clinician.
  CFS evaluates specific domains, including comorbidity, function, and cognition, to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill). A higher score indicates a higher illness.
Mean change from baseline in quality of life as measured by change in the Falls Efficacy Scale- International (FES-I) questionnaire score. | Day 0 (baseline), Week 6, 12, 24, 36, 52
  The Falls Efficacy Scale- International (FES-I) is a 16-item questionnaire that assesses concern about falling during daily activities.
  Scores range from 16 (no concern) to 64 (severe concern). A lower score indicates a lower fear of falling.
Mean change from baseline in quality of life as measured by change in the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 20a score. | Day 0 (baseline), Week 6, 12, 24, 36, 52
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 20a assesses one's ability to carry out activities that require physical actions, ranging from self-care (activities of daily living) to more complex activities that require a combination of skills, often within a social context.
  Subjects will rank 20 questions from a scale of 1 to 5, with 5 being the highest physical function and 1 being the lowest. The score will be added up, and the Raw score will be converted to T-Score using the PROMIS Adult v2.0 Physical Function 20a Short Form Conversion Table.
Mean change from baseline in quality of life as measured by change in the 36-Item Short Form survey (SF-36) score. | Day 0 (baseline), Week 6, 12, 24, 36, 52
  The 36-Item Short Form Survey (SF-36) is a patient-reported generic measure of health status. It consists of 36 items covering both mental and physical domains. Items include limitations in physical activities because of health problems, limitations in social activities because of physical or emotional problems, limitations in usual role activities because of physical health problems, bodily pain, general mental health (psychological distress and well-being), limitations in usual role activities because of emotional problems, vitality (energy and fatigue), and general health perceptions.

IPD SHARING:
Plan to Share IPD: No